CLINICAL TRIAL: NCT02601027
Title: A Phase III Study of Pre-operative Transversus Abdominis Plane Blocks Using the Nimbus Ambulatory Infusion System in Patients Undergoing Abdominal Free Flap-based Breast Reconstruction
Brief Title: Transversus Abdominis Plane Block in Microsurgical Breast Recon w/Abdominal Free Flap in Breast CA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gordon Kwanlyp Lee, Professor of Surgery (Plastic and Reconstructive Surgery), Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-34315; BRS0058 (Other: OnCore)
Record Dates: First submitted 2015-11-04; First posted 2015-11-10 (Estimated); Results first posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-08

CONDITIONS: Breast - Female
MeSH Terms: interventions — Dental Occlusion; Bupivacaine; Acetaminophen; Hydromorphone; Oxycodone; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 0.125% Bupivacaine (Experimental): 0.125% bupivacaine infusion via transversus abdominis plane (TAP) catheter
  Interventions: Procedure: Transversus Abdominis Plane (TAP) block; Device: Nimbus Infusion Pump IV Administration; Drug: Bupivacaine infusion; Drug: Acetominophen; Drug: Hydromorphone; Drug: Oxycodone; Drug: Ondansetron
- Placebo (Placebo Comparator): Saline infusion (sham) via transversus abdominis plane (TAP) catheter.
  Interventions: Procedure: Transversus Abdominis Plane (TAP) block; Device: Nimbus Infusion Pump IV Administration; Drug: Acetominophen; Drug: Hydromorphone; Drug: Oxycodone; Drug: Ondansetron

INTERVENTIONS:
Procedure: Transversus Abdominis Plane (TAP) block
Device: Nimbus Infusion Pump IV Administration
Drug: Bupivacaine infusion
  Other Names: Exparel; Marcaine; Marcaine Spinal; Sensorcaine; Sensorcaine-MPF; Sensorcaine-MPF Spinal; ReadySharp bupivacaine; P-Care M
  Arms: 0.125% Bupivacaine
Drug: Acetominophen
  Other Names: Tylenol
Drug: Hydromorphone
  Other Names: Dilaudid; Dilaudid-HP; Exalgo
Drug: Oxycodone
  Other Names: Oxycontin; Xtampza ER; Oxaydo; Roxicodone
Drug: Ondansetron
  Other Names: Zofran; Zofran ODT; Zuplenz

SUMMARY:
The primary objective is to determine if pre-operative transversus abdominis plane (TAP) nerve blocks by continued infusion of local anesthetic post-operatively affects post-operative narcotic usage, as compared to a placebo TAP block, after breast reconstruction surgery.

DETAILED DESCRIPTION:
Primary Objective: The primary objective is to determine if pre-operative transversus abdominis plane (TAP) blocks with continued infusion of local anesthetic post-operatively affect post-operative narcotic usage as compared to a placebo TAP block.

Secondary Objectives:

* Determine if pre-operative TAP blocks with continued infusion of local anesthetic post-operatively affect post-operative pain scores as compared to a placebo TAP block.
* Determine if pre-operative TAP blocks with continued infusion of local anesthetic post-operatively affect anti-emetic usage as compared to a placebo TAP block.
* Determine if pre-operative TAP blocks with continued infusion of local anesthetic post-operatively affect time to ambulation post-operatively as compared to a placebo TAP block.
* Determine if pre-operative TAP blocks with continued infusion of local anesthetic post-operatively affect time to first bowel movement as compared to a placebo TAP block.
* Determine if pre-operative TAP blocks with continued infusion of local anesthetic post-operatively affect patient-reported quality of life as compared to a placebo TAP block.

ELIGIBILITY:
Inclusion Criteria

* Prior diagnosis or presumed diagnosis of breast cancer or undergoing prophylactic treatment.
* Greater than 18 years old.
* Female.
* Undergoing microsurgical breast reconstruction with abdominal free flap.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* True allergy to local anesthetics or opioids.
* History of addiction to narcotics within the last 24 months
* History of chronic pain on opioids within the last 24 months.
* Specific mental health issues such as schizophrenia or bipolar disorder.
* Patients who are pregnant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 120 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon K Lee, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mundy LR, Homa K, Klassen AF, Pusic AL, Kerrigan CL. Breast Cancer and Reconstruction: Normative Data for Interpreting the BREAST-Q. Plast Reconstr Surg. 2017 May;139(5):1046e-1055e. doi: 10.1097/PRS.0000000000003241. PMID 28445351
- [Background] Pusic AL, Klassen AF, Scott AM, Klok JA, Cordeiro PG, Cano SJ. Development of a new patient-reported outcome measure for breast surgery: the BREAST-Q. Plast Reconstr Surg. 2009 Aug;124(2):345-353. doi: 10.1097/PRS.0b013e3181aee807. PMID 19644246
- [Background] Voineskos SH, Klassen AF, Cano SJ, Pusic AL, Gibbons CJ. Giving Meaning to Differences in BREAST-Q Scores: Minimal Important Difference for Breast Reconstruction Patients. Plast Reconstr Surg. 2020 Jan;145(1):11e-20e. doi: 10.1097/PRS.0000000000006317. PMID 31577663
- [Result] Kwong JW, Tijerina JD, Choi S, Shakir A, Nguyen DH, Nazerali RS, Lee GK. Randomized Double-Blinded, Placebo-Controlled Trial: Transversus Abdominis Plane (TAP) Blocks in Breast Cancer Patients Undergoing Reconstruction with Abdominal Free Flap. Annual Meeting of the California Society of Plastic Surgeons. San Diego, California. May 19, 2018.

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.125% Bupivacaine: * 0.125% bupivacaine infusion through transversus abdominis plane (TAP) catheter
  * Transversus Abdominis Plane (TAP) block
  * Nimbus Infusion Pump IV Administration
  * Bupivacaine infusion
  * Acetominophen
  * Hydromorphone
  * Oxycodone
  * Ondansetron
- Placebo: * Saline infusion (sham) for transversus abdominis plane (TAP) catheter.
  * Transversus Abdominis Plane (TAP) block
  * Nimbus Infusion Pump IV Administration
  * Bupivacaine infusion
  * Acetominophen
  * Hydromorphone
  * Oxycodone
  * Ondansetron
Period: Registration to Surgery
Arm/Group | 0.125% Bupivacaine | Placebo
Started | 64 | 56
Completed | 44 | 46
Not Completed | 20 | 10
Not completed — Withdrawal by Subject | 20 | 10
Period: Surgery to Assessments
Arm/Group | 0.125% Bupivacaine | Placebo
Started | 44 | 46
Completed | 44 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 0.125% Bupivacaine: 0.125% bupivacaine infusion via transversus abdominis plane (TAP) catheter
  Transversus Abdominis Plane (TAP) block
  Nimbus Infusion Pump IV Administration
  Bupivacaine infusion
  Acetominophen
  Hydromorphone
  Oxycodone
  Ondansetron
- Placebo: Saline infusion (sham) via transversus abdominis plane (TAP) catheter.
  Transversus Abdominis Plane (TAP) block
  Nimbus Infusion Pump IV Administration
  Acetominophen
  Hydromorphone
  Oxycodone
  Ondansetron
- Total: Total of all reporting groups
Arm/Group | 0.125% Bupivacaine | Placebo | Total
Number analyzed (Participants) | 64 | 56 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 49 | 107
  >=65 years | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.24 (9.58) | 52.11 (10.50) | 51.11 (9.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 56 | 120
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 2 | 5
  White | 44 | 38 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 64 | 56 | 120

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Narcotic Usage
Description: Narcotic usage was collected for first 48 hours post-operatively after breast reconstruction. The type and amount of each narcotic administered were each converted to the morphine equivalent amount that would be orally administered to achieve the same event. This term is known as the oral morphine equivalent (OME). Narcotic usage was assessed between the group receiving transversus abdominis plane (TAP) nerve block compared to the group receiving the placebo control. The outcome is reported as the observed OME for each group.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 46
milligrams (mg) | 139.3 (117.2) | 169.2 (136.5)

2. Secondary Outcome: Post-operative Pain Score
Description: Post-operative Pain Score is defined using Visual Analog Scale (VAS), a patient-reported pain score based on viewing a graphic of a scale 0 to 10, and indicating pain level. Each participant was asked about 48 hours after breast reconstruction to indicate their their perceived pain according on the VAS scale. Higher scores represent greater pain. The outcome is reported as the mean VAS score at 48 hours, with standard deviation.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 46
units on a scale | 3.76 (1.72) | 3.96 (2.14)

3. Secondary Outcome: Post-operative Anti-emetic Usage
Description: Odansetron by intravenous administration was used to control nausea (ie, an anti-emetic drug). Anti-emetic usage was collected for first 48 hours post-operatively after breast reconstruction for the group receiving transversus abdominis plane (TAP) nerve block compared to the group receiving the placebo control. The outcome is reported as the mean quantity of Odansetron in milligrams (mg) administered to each group, with standard deviation.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 46
milligrams (mg) | 5.14 (5.30) | 9.93 (13.74)

4. Secondary Outcome: Time to Ambulation
Description: Time to ambulation is defined as the amount of time, from midnight on post-operative Day 1 (ie, first midnight following the surgery), to when the participant to be able to stand up and walk a few steps post-operatively. The assessment of whether or not the participant was able to walk was subjective on the part of the shift nurse (ie, no defined number of steps nor quantitative assessment of gait or stability), and was not explicitly defined in the protocol or elsewhere. The outcome is reported as the time to ambulation in days, with standard deviation, for the group receiving transversus abdominis plane (TAP) nerve block and the group receiving the placebo control.
Time Frame: up to 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 46
days | 1.28 (0.52) | 1.45 (0.62)

5. Secondary Outcome: Time to First Bowel Movement
Description: Time to first bowel movement is defined as the amount of time, from midnight on post-operative Day 1 (ie, first midnight following the surgery), to when the participant was to be able to pass a stool post-operatively. The outcome is reported as the time in days, with standard deviation, for the group receiving transversus abdominis plane (TAP) nerve block and the group receiving the placebo control.
Time Frame: up to 1 week
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 44 | 46
days | 1.67 (1.08) | 1.62 (0.99)

6. Secondary Outcome: Quality of Life Measurement
Description: Quality of life for the study groups was assessed with the BREAST-Q questionnaire, a survey set of 6 pre-operative questionnaires comprised of 58 questions, and 15 post-operative questionnaires, collected 2 to 6 months after surgery, which is comprised of 109 questions. The results range for the pre-operative and post-operative questionnaire sets is 0 to 269 and 0 to 462, respectively. Because the baseline and post-operative domains are different, the BREAST-Q survey is not a measure of quality of life change over time. The Breast Q questionnaire was validated by Pusic, et al (citation provided). Higher scores for a domain represents better quality of life. The outcome is reported as the mean for each group and timepoint, with standard deviation.
Time Frame: Pre-operative Baseline and Post-operative (2-6 months)
Population: Most participants were lost to follow-up, and did not return the case report form (CRF) for this patient-reported Quality of Life (QoL) data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.125% Bupivacaine | Placebo
Number analyzed (Participants) | 10 | 7
score on a scale
  Pre-operative baseline | 97.30 (17.61) | 99.08 (20.73)
  Post-operative (2 to 6 month) | 342.11 (26.42) | 358.00 (16.83)

ADVERSE EVENTS:
Time Frame: Through 7 days post-operative
Arm/Group | 0.125% Bupivacaine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/56
Other Adverse Events (participants affected / at risk) | 21/64 | 27/56
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.125% Bupivacaine (N=64) | Placebo (N=56)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Chest wall necrosis, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (2)
Localized Edema (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT02601027/Prot_SAP_000.pdf